CLINICAL TRIAL: NCT02239952
Title: Pilot Study on the Determination of Tumor Concentrations of Protein Kinase Inhibitors in Patients With Newly Diagnosed High-grade Glioma
Brief Title: HGG-TCP (High Grade Glioma - Tumor Concentrations of Protein Kinase Inhibitors)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.E. van Linde, Medical Oncologist, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.465
Record Dates: First submitted 2014-08-28; First posted 2014-09-15 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cancer; High-grade Glioma
MeSH Terms: conditions — Neoplasms; Glioma | interventions — Sunitinib; vandetanib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sunitinib (Experimental)
  Interventions: Drug: Sunitinib
- vandetanib (Experimental)
  Interventions: Drug: vandetanib
- Erlotinib (Experimental)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Sunitinib — 50 mg once daily, oral use for 14 days
  Arms: sunitinib
Drug: vandetanib — 300 mg, once daily, oral use for 14 days
  Arms: vandetanib
Drug: Erlotinib — 150 mg, once daily, oral use for 14 days
  Arms: Erlotinib

SUMMARY:
The purpose of this study is to determine intratumoral concentration of kinase inhibitors upon 2 weeks of treatment in tumor tissue (in the brain) of patients with high-grade gliomas (HGG).

DETAILED DESCRIPTION:
In clinical trials for HGG, multiple agents targeting various oncogenic signaling pathways that play an important role in the biology of HGG have been studied, but unfortunately only a small number of patients seem to benefit from these treatment strategies. Whether these disappointing results are due to a restricted drug delivery through the blood-brain barrier, or due to differential biological characteristics of these HGGs, remains unknown. To better understand these clinical observations and to find potential insight how to overcome them, we intend to measure tumor concentrations of PKIs after approximately two weeks treatment and to determine whether these tumor concentrations correlate with plasma- and CSF concentrations of PKIs. Subsequently, we intend to determine the (phospho)proteomic profiles and kinase inhibitory activity in tumor tissue from these HGG patients after approximately two weeks of treatment with a PKI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients without a history of brain tumor
2. Initial brain MR-scan suggesting a high grade glioma, according to the interpretation of an expert neuroradiologist
3. On initial MR-scan a tumor localisation that is deemed resectable without major neurological deficits
4. Patients must have a Karnofsky Performance Score ≥ 70%
5. Patients must have a RTOG Neurologic Function Status of 0-2
6. Patients need to have adequate hematological, renal and hepatic function as assessed by the following laboratory requirements to be conducted within seven days prior to start study treatment: - Hemoglobin > 7.0 mmol/l - Absolute neutrophil count (ANC) >1,5 x 10*9/l - Platelet count > 100 x 10*9/l - ALT and AST< 2.5 x ULN - Alkaline phosphatase < 4 x ULN - Serum creatinine eGFR > 50 ml/min
7. Patients are 18 years of older
8. Male and female patients with reproductive potential must use an approved contraceptive method during and for three months after discontinuation of study treatment
9. Patients need to give informed consent
10. Patients should be able to swallow oral medication

Exclusion Criteria:

1. Patients receiving prior chemotherapy, radiotherapy or anti-angiogenic therapy
2. Use of anti-coagulant therapy
3. Use of CYP3A4 enzyme-inducing drugs, other than dexamethasone (including Carbamazepine, Phenytoine, Phenobarbital)
4. Initial MR-scan of the brain showing tumor hemorrhage or intracerebral hemorrhage
5. Patients with progressive neurological symptoms despite dexamethasone
6. Inability to comply with protocol or study procedures
7. Pregnancy
8. Patients with uncontrolled arterial hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen.
9. Patients with a history of cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
10. Patients with evidence or history of bleeding diathesis
11. Patients with a history of venous or arterial thrombo-embolic events or hemorrhagic disease during the past six months
12. Patients with a history of congestive heart failure (NYHA III, IV)
13. Patients with a history of peripheral vascular disease (Fontaine stage III and IV)
14. Patients with stroke or myocardial infarction during the past six months
15. Patients with a history of a recent peptic ulcer disease (endoscopically-proven gastric ulcer, duodenal ulcer of esophageal ulcer) during the past six months
16. Patients with uncontrolled infections (> grade 2 NCI-CTC version 4.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
PKI and active metabolites concentrations in tumor tissue | 2 weeks
  PKI concentrations and active metabolites in tumor tissue after approximately two weeks of PKI treatment will be determined.

SECONDARY OUTCOMES:
Correlation of PKI and active metabolites concentrations in tumor. | 2 weeks
  Venous blood sampling will be performed to determine plasma drug and active metabolites concentrations after approximately one and two weeks of PKI treatment and during surgery. CSF samples will be drawn during surgery. Plasma- and CSF drug concentrations will be correlated to tumor drug concentrations. Plasma samples for pharmacodynamics will be simultaneously drawn with the on- and after treatment hematology and chemistry analysis.
Feasibility of determining the (phospho)proteomic profiles and kinase activity profiles in tumor tissue and CSF. | 2 weeks
  Kinome wide and quantitative (phospho)proteomic profiles will be determined in tumor tissue of study patients and in tumor tissue of matched controled patients. We anticipate that these profiles will reveal information on the effect of treatment on kinase abundances, phosphopeptide levels and on phosphorylation sites. Differences in levels of phosphopeptides and fold-change of phosphorylation sites will be quantified. In an exploratory design, we will determine whether observed profile differences can be correlated to drug concentrations in tumor tissue. Kinase inhibition profiles will be measured according to standard methods as developed and modified in our laboratory.
Significant difference of the (phospho)proteomic profiles and kinase activities of tumor tissue in study patients and control group. | 2 weeks
  The (phospho)proteomic profiles and kinase activity profiles will be determined in tumor tissue of study patients and in tumor tissue of patients in a control group.
  Kinase inhibition profiles will be measured according to standard methods as developed and modified in our laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Linde ME, Labots M, Brahm CG, Hovinga KE, De Witt Hamer PC, Honeywell RJ, de Goeij-de Haas R, Henneman AA, Knol JC, Peters GJ, Dekker H, Piersma SR, Pham TV, Vandertop WP, Jimenez CR, Verheul HMW. Tumor Drug Concentration and Phosphoproteomic Profiles After Two Weeks of Treatment With Sunitinib in Patients with Newly Diagnosed Glioblastoma. Clin Cancer Res. 2022 Apr 14;28(8):1595-1602. doi: 10.1158/1078-0432.CCR-21-1933. PMID 35165100